CLINICAL TRIAL: NCT00811291
Title: SIMBA-Study Investigating Mental Acuity Effects of B-vitamins in Children
Brief Title: Influence of Vitamin-B-complex on Cognitive Ability of Kindergarten Kids
Acronym: SIMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: European Union (Other); Unilever R&D (Industry)
Responsible Party: Principal Investigator, Koletzko - Office, Professor Berthold Koletzko, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08032V
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: B-vitamins; Folic-Acid; kindergarten kids; cognitive tests; Healthy kids; second part low urine vitamine-B-metabolites
MeSH Terms: interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Dietary Supplement: calcium
- 2 (Active Comparator): folic acid and B-vitamin supplement
  Interventions: Dietary Supplement: Vitamine-B and Folic Acid Complex, calcium

INTERVENTIONS:
Dietary Supplement: Vitamine-B and Folic Acid Complex, calcium — 90 days of intake, will be given in drink (e.g. tea, milk, juice). Dosage within official recommendations for kindergarten kids
  Arms: 2
Dietary Supplement: calcium — according to protocol
  Arms: 1

SUMMARY:
Vitamin-B and Folic intake of Kindergarten kids in Germany is only 50-70% of the official recommendations. In studies with adults it has been found that for example providing people suffering from Alzheimer´s disease improved their mental and cognitive abilities when provided with a high intake of these vitamins.The hypothesis is, that kindergarten kids, 4-6 years of age, could also improve mentally from a recommended intake of B-vitamins and Folic Acid.

1. screening study: The urine of 1200 kindergarten kids will be analyzed for metabolites of these vitamins, and the 250 kids with the lowest results will be invited for a randomized double blind intervention study.
2. intervention study: Participating kids will get an one hour mental and cognitive testing before and after the intervention. The intervention will be one portion of the recommended dosage of a vitamin B complex and folic acid , given in a drink (milk, tea, etc). The assumption is, that the treatment group will perform better than the placebo group in the second test phase.

ELIGIBILITY:
Inclusion Criteria:

* age: 4-6 years
* kindergarten kids in Munich
* fluent in German
* healthy
* no medication

Exclusion Criteria:

* not fluent in German
* chronic illness
* intake of multivitamin supplements

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in outcome of cognitive testing of kindergarten kids after intervention | August 2009

SECONDARY OUTCOMES:
Analysis of Vitamine-B-metabolites in urine of kindergarten kids via a new method | September 2008-December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Berthold V Koletzko, M.D., PhD, Principal Investigator — Dr. von Hauner Children´s Hospital, Ludwig-Maximilians-University, Munich
Locations (1):
- Dr. von Hauner Children´s Hospital, Munich, Germany